CLINICAL TRIAL: NCT05003817
Title: Controlled Trial of High-risk Coronary Intervention With Percutaneous Left Ventricular Unloading
Acronym: CHIP-BCIS3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); The Queen Elizabeth Hospital (Other); The Royal Bournemouth Hospital (Other); St. George's Hospital, London (Other); King's College Hospital NHS Trust (Other); King's College London (Other); Royal Victoria Hospital, Belfast (Other); Bristol Heart Institute (Unknown); Barts Heart Centre, London (Unknown); Glenfield Hospital, Leicester (Other); Morriston Hospital, Swansea (Unknown); St Thomas' Hospital, London (Other); New Cross Hospital, Wolverhampton (Unknown); Essex Cardiothoracic Centre, Basildon (Unknown); Freeman Hospital, Newcastle (Unknown); Golden Jubilee National Hospital, Glasgow (Unknown); John Radcliffe Hospital, Oxford (Unknown); Manchester Royal Infirmary (Unknown); Royal Cornwall Hospital, Truro (Unknown); Royal Brompton & Harefield NHS Foundation Trust (Other); Musgrove Park Hospital, Taunton (Unknown); Royal Sussex County Hospital, Brighton (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS290599; 130593 (Other Grant/Funding Number: NIHR HTA CET); 17730734 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2021-07-21; First posted 2021-08-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease
Keywords: percutaneous coronary intervention; percutaneous left ventricular unloading
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LV-unloading (Experimental): Participants in the elective unloading (intervention) group will have a percutaneous left ventricular unloading device (pLVAD) inserted at the start of the procedure, before the coronary intervention. Maximal support will be provided throughout the procedure, following which support will be weaned and the device removed should the patient remain haemodynamically stable.
  Interventions: Device: Percutaneous left ventricular unloading
- Standard of Care (No Intervention): Participants in the control arm will receive the planned high-risk percutaneous coronary intervention as is the current standard of care without elective left ventricular unloading. Alternative mechanical circulatory support devices (such as the intra-aortic balloon pump (IABP) or extracorporeal membrane oxygenation (ECMO) will only be permitted in case of complications.

INTERVENTIONS:
Device: Percutaneous left ventricular unloading — Percutaneous left ventricular unloading involves the placement of a mechanical pump which draws blood from the left ventricle and returns it into the aorta at flow rates approaching native cardiac output.
  Arms: LV-unloading

SUMMARY:
Over 100,000 coronary stent procedures, where small balloons are used to stretch open a narrowed blood vessel, are performed every year in the United Kingdom to treat people who have conditions such as angina or have suffered a heart attack.

For most patients the risk of complications is low, but for some, there is a higher risk of their heart failing during the procedure. Heart failure is a serious complication which can need treatment with a life support machine and lead to major damage to the heart muscle or even death. These risks are greatest in patients with severely diseased heart arteries and those who already have weakened heart muscle.

A new technology may be able to help with this problem. It consists of a small heart pump which is placed in the heart's main pumping chamber (the left ventricle, LV). This pump is known as a LV unloading device. The LV unloading device is inserted into the heart through a blood vessel in the leg and supports the heart muscle. It is removed at the end of the procedure or when the heart can pump safely on its own. Whilst this heart pump is promising, it comes with some risks of its own. These include bleeding and damage to the arteries in the legs. It is also expensive, costing £8,000 per operation. Currently, there is no strong evidence to guide the use of this device.

The CHIP-BCIS3 study aims to determine whether these heart pumps are beneficial and cost-effective in patients receiving a stenting procedure who are at high-risk of complications.

ELIGIBILITY:
Inclusion Criteria:

1. Extensive coronary disease defined by a British Cardiovascular Intervention Society (BCIS) Jeopardy Score ≥ 8*
2. Severe left ventricular systolic dysfunction defined as a LVEF ≤ 35% (or ≤ 45% in the presence of severe mitral regurgitation)#
3. Complex PCI defined by the presence of at least one of the following criteria:

   * Unprotected left main intervention in the presence of

     * an occluded dominant right coronary artery, or
     * a left dominant circulation, or
     * disease involving the entire bifurcation (Medina 1,1,1 or 0,1,1)
   * Intended calcium modification (by rotational or orbital atherectomy, lithotripsy or laser)

     * in multiple vessels or
     * in the left main stem, or
     * in a final patent conduit, or
     * where the anatomic SYNTAX score is ≥32
   * Target vessel is a chronic total occlusion with planned retrograde approach

     * In general, patients who do not have bypass grafts will be eligible if the patient has at least proximal left anterior descending (LAD) disease or at least proximal 2 vessel disease. For patients with patent bypass grafts, or in cases where the extent of coronary artery disease (CAD) is uncertain, the BCIS-1 JS should be calculated. The maximum possible JS score is 12. N.B. The JS should be based on all coronary disease, not just the vessel subtending viable myocardium.

       * Biplane / 3D echocardiography, or cardiac MRI can be used to assess the qualifying LVEF.

Exclusion Criteria:

1. Cardiogenic shock or acute STEMI at randomisation (including current treatment with a mechanical circulatory support device)
2. Contraindication to pLVAD insertion
3. Inability to give informed consent
4. Previously enrolled in CHIP or current enrolment in another interventional study that may affect CHIP outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite hierarchical outcome analysed using a Win Ratio method. | Minimum 12-months of follow-up, up to 51 months
  Events included in the composite hierarchical outcome include: death, stroke, spontaneous myocardial infarction, cardiovascular hospitalisation or periprocedural myocardial infarction.

SECONDARY OUTCOMES:
Individual components of the primary outcome including: death, stroke, spontaneous myocardial infarction, cardiovascular hospitalisation or periprocedural myocardial injury. | Minimum 12-months of follow-up, up to 51 months
  Analysis will include repeated occurrences of these events
Completeness of revascularisation measured by the change in anatomic BCIS-JS score | Between baseline and the completion of the final planned PCI procedure, up to a maximum of 1 year
Completeness of revascularisation measured by the change in anatomic SYNTAX score | Between baseline and the completion of the final planned PCI procedure, up to a maximum of 1 year
Major bleeding using the Bleeding Academic Research Consortium (BARC 3 to 5) classification | At 90 days, 1, 2, 3 and 4 years post-randomisation, up to a maximum of 51 months of follow-up
Vascular complication measured using VARC criteria | Post-procedural at each planned percutaneous coronary intervention procedure, up to a maximum of 1 year
Procedural complication measured as the incidence of VT/VF requiring defibrillation, cardiorespiratory arrest, acute pulmonary oedema requiring assisted ventilation or prolonged hypotension | Post-procedural at each planned percutaneous coronary intervention procedure, up to a maximum of 1 year
Unplanned revascularisation | At 90 days, 1, 2, 3 and 4 years post-randomisation, up to a maximum of 51 months of follow-up
Health-related quality of life and functional status measured by the EuroQol 5-Dimension 5-level questionnaire (EQ-5D- 5L) | At 90 days, 1, 2, 3 and 4 years post-randomisation, up to a maximum of 51 months of follow-up
  The EuroQol 5-Dimension 5-level questionnaire (EQ-5D- 5L) measures quality of life and functional status with higher scores indicating better outcomes.
Resource utilisation and cost effectiveness measured by incremental costs | At 12-months post-randomisation
Resource utilisation and cost effectiveness measured by quality-adjusted life years (QALYs) | At 12-months post-randomisation
Resource utilisation and cost effectiveness measured by net monetary benefit | At 12-months post-randomisation
Acute kidney injury | At 90 days post-randomisation
  Defined as prolongation hospital admission or readmission ≥ 24 hours with rise in creatinine to 200% of baseline value or need for new renal replacement therapy within 30 days of procedure
Serial cardiac troponin (T or I) levels | At baseline, 6 and 24 hours post-procedure
  Measured by immunoassay
Length of stay | Up to a maximum of 1 year
  Measured by the duration of admission in complete days following the index PCI procedure and any subsequent planned staged PCI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Divaka Perera, Principal Investigator — KCL, GSTT
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ryan M, Ezad SM, Webb I, O'Kane PD, Dodd M, Evans R, Laidlaw L, Khan SQ, Weerackody R, Bagnall A, Panoulas VF, Rahman H, Strange JW, Fath-Ordoubadi F, Hoole SP, Stables RH, Curzen N, Clayton T, Perera D; CHIP-BCIS3 Investigators. Percutaneous Left Ventricular Unloading During High-Risk Coronary Intervention: Rationale and Design of the CHIP-BCIS3 Randomized Controlled Trial. Circ Cardiovasc Interv. 2024 Mar;17(3):e013367. doi: 10.1161/CIRCINTERVENTIONS.123.013367. Epub 2024 Feb 27. PMID 38410944

DOCUMENTS (1):
  • Study Protocol (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT05003817/Prot_000.pdf